CLINICAL TRIAL: NCT02948517
Title: Time Restricted Feeding for Weight Loss and Cardio-protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20160119
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Coronary Disease; Weight Loss
MeSH Terms: conditions — Coronary Disease; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Time restricted feeding (Experimental): Time restricted feeding
  Interventions: Other: Time restricted feeding
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Time restricted feeding — Time restricted feeding
  Arms: Time restricted feeding

SUMMARY:
Time restricted feeding (TRF) is a novel form of intermittent fasting that involves confining the period of food intake to 8 h/d (e.g. 10 am to 6 pm) without calorie counting. TRF is effective for weight loss and cardio-protection in obese adults. It is of great interest to see whether subjects can adhere to TRF for longer periods of time, and to see what degree of weight loss that can be achieved with TRF. Accordingly, the aims of this trial are: Aim 1: To determine if TRF can be implemented to facilitate weight loss in obese adults, and Aim 2: To determine if TRF can produce clinically meaningful reductions in plasma lipids, blood pressure, insulin resistance, and inflammatory markers.

DETAILED DESCRIPTION:
Time restricted feeding (TRF) is a novel form of intermittent fasting that involves confining the period of food intake to 8 h/d (e.g. 10 am to 6 pm) without calorie counting. Recent findings from short-term uncontrolled trials suggest that TRF is effective for weight loss and cardio-protection in obese adults. In view of these pilot findings, it is of great interest to see whether subjects can adhere to TRF for longer periods of time, and to see what degree of weight loss that can be achieved with TRF. Accordingly, the aims of this trial are: Aim 1: To determine if TRF can be implemented to facilitate weight loss in obese adults, and Aim 2: To determine if TRF can produce clinically meaningful reductions in plasma lipids, blood pressure, insulin resistance, and inflammatory markers. To test the study objectives, a 14-week randomized, controlled, parallel-arm trial, divided into 2 consecutive periods: (1) 2-week baseline; and (2) 12-week weight loss, will be implemented. Obese subjects (n = 40) will be randomized to 1 of 2 groups: (1) TRF (n = 20), or (2) control (n = 20). This study will be the first randomized controlled trial of TRF, and will show that TRF can be implemented to help obese individuals lose weight and lower risk of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Body mass index (BMI) between 30.0 and 40 kg/m2
* Age between 25 and 65 years
* Sedentary (light exercise less than 1 h per week) or moderately active (moderate exercise 1 to 2 h per week)
* Weight stable for >3 months prior to the beginning of the study (gain or loss <4 kg)
* Able to give written informed consent

Exclusion Criteria:

* Smoker
* Diabetic
* History of cardiovascular disease (myocardial infarction or stroke)
* Taking weight loss medications
* History of eating disorders
* Night-shift workers
* Perimenopausal
* Pregnant or trying to become pregnant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks

SECONDARY OUTCOMES:
Plasma lipids | 12 weeks
Blood pressure | 12 weeks
Insulin resistance measured by Homeostatic model assessment (HOMA) | 12 weeks
Inflammatory markers: Tumor necrosis factor-alpha (TNF) and Interleukin-6 (IL-6) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717